CLINICAL TRIAL: NCT01720290
Title: A 3-month, Open-label, Randomized, Multi-center Study of Repaglinide in Combination With Metformin as Compared to Metformin or Repaglinide Given as Monotherapy for the Treatment of Type 2 Diabetes.
Brief Title: Comparison of Repaglinide and Metformin Administered Alone or in Combination in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-3018
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rep (Experimental)
  Interventions: Drug: repaglinide
- Met (Active Comparator)
  Interventions: Drug: metformin
- Rep + met (Active Comparator)
  Interventions: Drug: repaglinide; Drug: metformin

INTERVENTIONS:
Drug: repaglinide — Dose individually adjusted
  Arms: Rep; Rep + met
Drug: metformin — Dose individually adjusted
  Arms: Met
Drug: metformin — Dose at 1000 mg/day
  Arms: Rep + met

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare repaglinide and metformin administered alone or in combination in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated with oral hypoglycaemic agents (OHA) as monotherapy (if metformin, less than 1500 mg daily)
* Body Mass Index (BMI) of 21-35 kg/m^2
* HbA1c (glycosylated haemoglobin A1c) between 7.0-10%

Exclusion Criteria:

* Treatment with insulin within the last 3 months preceding the trial
* Uncontrolled treated or untreated hypertension (systolic blood pressure above or equal to 180 mm Hg, and/or diastolic blood pressure above 105 mm Hg)
* Participation in any other clinical trial within 30 days of screening

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-07-25 (Actual); Primary Completion 2003-02-25 (Actual); Study Completion 2003-02-25 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin A1c)

SECONDARY OUTCOMES:
Fasting blood glucose (FBG)
1-hour post prandial blood glucose (PPBG)
Incidence of hypoglycemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- China (3):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Beijing
  - Novo Nordisk Investigational Site, Shanghai

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com